CLINICAL TRIAL: NCT01407861
Title: Aerobic Endurance Training Versus Relaxation Training in Migraine Prophylaxis
Brief Title: Aerobic Endurance Training vs. Relaxation Training in Patients With Migraine
Acronym: ARMIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Hans-Christoph Diener, Prof. of Neurology, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aerobic-Relax-Migraine
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation training (Active Comparator): Patients participate in a relaxation training program under expert guidance at least three times a week over 12 weeks.
  Interventions: Other: Relaxation Training
- Aerobic endurance training (Active Comparator): Patients participate in a moderate aerobic endurance training program under expert guidance three times a week over 12 weeks.
  Interventions: Other: Aerobic endurance Training

INTERVENTIONS:
Other: Relaxation Training — Patients participate in a relaxation training program under expert guidance at least three times a week over 12 weeks.
  Arms: Relaxation training
Other: Aerobic endurance Training — Patients participate in a moderate aerobic endurance training program under expert guidance three times a week over 12 weeks.
  Arms: Aerobic endurance training

SUMMARY:
This is a single centre, open label, prospective, randomized study on the prophylactic effect of moderate aerobic endurance training versus relaxation training in patients with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Patient's signature on the informed consent document [each patient should be given ample time to read (or have read to them) the consent form, ask any questions they may have regarding the trial and have a clear understanding of the trial and the procedures involved prior to the signing of the consent form].
* Patients have a clinical diagnosis of migraine with or without aura according to IHS criteria at least one year prior to enrollment.
* Patients have a clinical diagnosis of migraine with or without aura and in addition a clinical diagnosis of tension type headache according to IHS criteria, if patients are able to differentiate between the two headache diagnoses and if migraine is more frequent in these patients
* Patients that report at least three headache days per month

Exclusion Criteria:

* Diseases or disabilities that disqualify to perform either aerobic endurance training or relaxation training
* Language difficulties that disable to fill out questionnaires
* Pregnancy
* Additional diagnosis of secondary headache according to the IHS criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reduction of headache days in the last 4 weeks of the 12-week training compared to baseline (4 weeks before start of the training). | 16 weeks

SECONDARY OUTCOMES:
Number of headache days 12 weeks after finishing the training (follow up). | 20 weeks
Consumption of analgetic agents/triptans | 20 weeks
Increase in aerobic capability | 12 weeks
Impact on burden of disease | 20 weeks
Psychological Impact of Training | 20

CONTACTS AND LOCATIONS:
Overall Officials: Charly Gaul, MD, Principal Investigator — Department of Neurology, University of Duisburg-Essen
Locations (1):
- Department of Neurology, University of Duisburg-Essen, Essen, Germany

REFERENCES:
- [Derived] Totzeck A, Unverzagt S, Bak M, Augst P, Diener HC, Gaul C. Aerobic endurance training versus relaxation training in patients with migraine (ARMIG): study protocol for a randomized controlled trial. Trials. 2012 Apr 27;13:46. doi: 10.1186/1745-6215-13-46. PMID 22540391